CLINICAL TRIAL: NCT00318461
Title: Liraglutide Effect and Action in Diabetes (LEAD-2): Effect on Glycaemic Control After Once Daily Administration of Liraglutide in Combination With Metformin Versus Metformin Monotherapy Versus Metformin and Glimepiride Combination Therapy in Subjects With Type 2 Diabetes
Brief Title: To Compare the Effect of Liraglutide When Given Together With Metformin With the Effect of Metformin Given Alone and With the Effect of Glimepiride and Metformin Given Together
Acronym: LEAD-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1572
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Results first posted 2010-03-12 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lira 0.6 + Met (Experimental): Liraglutide 0.6 mg/day + glimepiride placebo + metformin 1.5-2.0 g/day
  Interventions: Drug: liraglutide; Drug: metformin; Drug: placebo
- Lira 1.2 + Met (Experimental): Liraglutide 1.2 mg/day + glimepiride placebo + metformin 1.5-2.0 g/day
  Interventions: Drug: metformin; Drug: placebo; Drug: liraglutide
- Lira 1.8 + Met (Experimental): Liraglutide 1.8 mg/day + glimepiride placebo + metformin 1.5-2.0 g/day
  Interventions: Drug: metformin; Drug: placebo; Drug: liraglutide
- Met Mono (Active Comparator): Metformin 1.5-2.0 g/day + liraglutide placebo + glimepiride placebo
  Interventions: Drug: metformin; Drug: placebo
- Met + Glim (Active Comparator): Glimepiride 4 mg/day + metformin 1.5-2.0 g/day + liraglutide placebo
  Interventions: Drug: metformin; Drug: glimepiride; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 0.6 mg for s.c. (under the skin) injection.
  Arms: Lira 0.6 + Met
Drug: metformin — 1.5-2.0 g tablets
Drug: glimepiride — 4 mg tablets
  Arms: Met + Glim
Drug: placebo — Glimepiride placebo 1 mg and 2 mg tablets
  Arms: Lira 0.6 + Met; Lira 1.2 + Met; Lira 1.8 + Met; Met Mono
Drug: placebo — Liraglutide placebo 1-3 mL for s.c. (under the skin) injection
  Arms: Met + Glim; Met Mono
Drug: liraglutide — 1.2 mg for s.c. (under the skin) injection
  Arms: Lira 1.2 + Met
Drug: liraglutide — 1.8 mg for s.c. (under the skin) injection
  Arms: Lira 1.8 + Met

SUMMARY:
This trial is conducted in Europe, Oceania, Africa, Asia and South America. This trial is designed to show the effect of treatment with liraglutide when adding to existing metformin therapy and to compare it with the effects of metformin monotherapy and combination therapy of metformin and glimepiride. Two trial periods: A 6 month (26 weeks) randomised, double-blinded period followed by an 18 months open-label extension, in total 2 years (104 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 2 diabetes and treated with oral anti-diabetic drugs (OADs) for at least 3 months
* HbA1c: 7.0-11.0 % (both incl.) in subjects on OAD monotherapy. 7.0-10.0 % (both incl.) in subjects on OAD combination therapy
* Body Mass Index (BMI) less than or equal 40 kg/m2

Exclusion Criteria:

* Subjects treated with insulin within the last three months
* Subjects with any serious medical condition
* Females of child bearing potential who are pregnant, breast-feeding or have the intention of becoming pregnant or not using adequate contraceptive methods
* Subjects using any drug (except for OADs), which in the Investigator's opinion could interfere with the glucose level (e.g. systemic corticosteroids)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1091 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (171):
- Argentina (4):
  - Novo Nordisk Investigational Site, Ciudad Autonoma de Bs As
  - Novo Nordisk Investigational Site, Ciudad Autónoma de Bs As
  - Novo Nordisk Investigational Site, Ciudad Autónoma de BsAs
  - Novo Nordisk Investigational Site, Junín
- Australia (21):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Penrith, New South Wales
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Daw Park, South Australia
  - Novo Nordisk Investigational Site, East Ringwood, Victoria
  - Novo Nordisk Investigational Site, Fremantle, Western Australia
  - Novo Nordisk Investigational Site, Adelaide
  - Novo Nordisk Investigational Site, Auckland
  - Novo Nordisk Investigational Site, Bankstown
  - Novo Nordisk Investigational Site, Box Hill
  - Novo Nordisk Investigational Site, Cairns
  - Novo Nordisk Investigational Site, Camperdown
  - Novo Nordisk Investigational Site, Christchurch
  - Novo Nordisk Investigational Site, Clayton
  - Novo Nordisk Investigational Site, Fitzroy
  - Novo Nordisk Investigational Site, Garran
  - Novo Nordisk Investigational Site, Hornsby
  - Novo Nordisk Investigational Site, Malvern
  - Novo Nordisk Investigational Site, Perth
  - Novo Nordisk Investigational Site, Westmead
  - Novo Nordisk Investigational Site, Woodville
- Belgium (6):
  - Novo Nordisk Investigational Site, Arlon
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Huy
  - Novo Nordisk Investigational Site, La Louvière
  - Novo Nordisk Investigational Site, Leuven
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Denmark (10):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Frederiksberg
  - Novo Nordisk Investigational Site, Herlev
  - Novo Nordisk Investigational Site, Hjørring
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, København S
  - Novo Nordisk Investigational Site, Odense
  - Novo Nordisk Investigational Site, Viborg
- Germany (38):
  - Novo Nordisk Investigational Site, Aschaffenburg
  - Novo Nordisk Investigational Site, Bad Heilbrunn
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Lauterberg im Harz
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Bad Neuenahr-Ahrweiler
  - Novo Nordisk Investigational Site, Beckum
  - Novo Nordisk Investigational Site, Bensheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Cologne
  - Novo Nordisk Investigational Site, Darmstadt
  - Novo Nordisk Investigational Site, Diez
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Flensburg
  - Novo Nordisk Investigational Site, Großheirath
  - Novo Nordisk Investigational Site, Halle
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Kutenholz-Mulsum
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Oberhausen
  - Novo Nordisk Investigational Site, Pirna
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Regensburg
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saaldorf
  - Novo Nordisk Investigational Site, Saarbrücken
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Speyer
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Sulzbach-Rosenberg
  - Novo Nordisk Investigational Site, Tübingen
  - Novo Nordisk Investigational Site, Viersen
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Würzburg
- Hungary (7):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Nyíregyháza
  - Novo Nordisk Investigational Site, Pécs
  - Novo Nordisk Investigational Site, Szekszárd
  - Novo Nordisk Investigational Site, Zalaegerszeg
- India (5):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Bangalore
- Ireland (2):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Waterford
- Italy (13):
  - Novo Nordisk Investigational Site, Bari
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Monza
  - Novo Nordisk Investigational Site, Orbassano
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Rimini
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Sassari
  - Novo Nordisk Investigational Site, Torino
  - Novo Nordisk Investigational Site, Verona
- Netherlands (4):
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, Sliedrecht
- Norway (10):
  - Novo Nordisk Investigational Site, Bekkestua
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Gjøvik
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kongsberg
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Tromsø
  - Novo Nordisk Investigational Site, Trondheim
- Romania (3):
  - Novo Nordisk Investigational Site, Cluj-Napoca, Cluj
  - Novo Nordisk Investigational Site, Constanța
  - Novo Nordisk Investigational Site, Iași
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Moldava nad Bodvou
  - Novo Nordisk Investigational Site, Prešov
  - Novo Nordisk Investigational Site, Trenčín
- South Africa (4):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Benoni
- Spain (15):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Alcázar de San Juan
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Bilbao
  - Novo Nordisk Investigational Site, Cadiz
  - Novo Nordisk Investigational Site, Girona
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Mérida
  - Novo Nordisk Investigational Site, San Cristóbal de La Laguna
  - Novo Nordisk Investigational Site, San Juan
  - Novo Nordisk Investigational Site, Santa Cruz de Tenerife
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Seville
- Sweden (7):
  - Novo Nordisk Investigational Site, Falun
  - Novo Nordisk Investigational Site, Karlstad
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Umeå
- United Kingdom (13):
  - Novo Nordisk Investigational Site, Abergavenny
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Berkshire
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, East Horsley
  - Novo Nordisk Investigational Site, Frome
  - Novo Nordisk Investigational Site, Llanelli
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Sunbury-on-Thames

REFERENCES:
- [Result] Nauck M, Frid A, Hermansen K, Shah NS, Tankova T, Mitha IH, Zdravkovic M, During M, Matthews DR; LEAD-2 Study Group. Efficacy and safety comparison of liraglutide, glimepiride, and placebo, all in combination with metformin, in type 2 diabetes: the LEAD (liraglutide effect and action in diabetes)-2 study. Diabetes Care. 2009 Jan;32(1):84-90. doi: 10.2337/dc08-1355. Epub 2008 Oct 17. PMID 18931095
- [Result] Sullivan SD, Alfonso-Cristancho R, Conner C, Hammer M, Blonde L. Long-term outcomes in patients with type 2 diabetes receiving glimepiride combined with liraglutide or rosiglitazone. Cardiovasc Diabetol. 2009 Feb 26;8:12. doi: 10.1186/1475-2840-8-12. PMID 19245711
- [Result] Nauck M, Marre M. Adding liraglutide to oral antidiabetic drug monotherapy: efficacy and weight benefits. Postgrad Med. 2009 May;121(3):5-15. doi: 10.3810/pgm.2009.05.1997. PMID 19491535
- [Result] McGill JB. Insights from the Liraglutide Clinical Development Program--the Liraglutide Effect and Action in Diabetes (LEAD) studies. Postgrad Med. 2009 May;121(3):16-25. doi: 10.3810/pgm.2009.05.1998. PMID 19491536
- [Result] Blonde L, Russell-Jones D. The safety and efficacy of liraglutide with or without oral antidiabetic drug therapy in type 2 diabetes: an overview of the LEAD 1-5 studies. Diabetes Obes Metab. 2009 Dec;11 Suppl 3:26-34. doi: 10.1111/j.1463-1326.2009.01075.x. PMID 19878259
- [Result] Jendle J, Nauck MA, Matthews DR, Frid A, Hermansen K, During M, Zdravkovic M, Strauss BJ, Garber AJ; LEAD-2 and LEAD-3 Study Groups. Weight loss with liraglutide, a once-daily human glucagon-like peptide-1 analogue for type 2 diabetes treatment as monotherapy or added to metformin, is primarily as a result of a reduction in fat tissue. Diabetes Obes Metab. 2009 Dec;11(12):1163-72. doi: 10.1111/j.1463-1326.2009.01158.x. PMID 19930006
- [Result] Buse JB, Garber A, Rosenstock J, Schmidt WE, Brett JH, Videbaek N, Holst J, Nauck M. Liraglutide treatment is associated with a low frequency and magnitude of antibody formation with no apparent impact on glycemic response or increased frequency of adverse events: results from the Liraglutide Effect and Action in Diabetes (LEAD) trials. J Clin Endocrinol Metab. 2011 Jun;96(6):1695-702. doi: 10.1210/jc.2010-2822. Epub 2011 Mar 30. PMID 21450987
- [Result] Bode BW, Brett J, Falahati A, Pratley RE. Comparison of the efficacy and tolerability profile of liraglutide, a once-daily human GLP-1 analog, in patients with type 2 diabetes >/=65 and <65 years of age: a pooled analysis from phase III studies. Am J Geriatr Pharmacother. 2011 Dec;9(6):423-33. doi: 10.1016/j.amjopharm.2011.09.007. Epub 2011 Nov 4. PMID 22055210
- [Result] Henry RR, Buse JB, Sesti G, Davies MJ, Jensen KH, Brett J, Pratley RE. Efficacy of antihyperglycemic therapies and the influence of baseline hemoglobin A(1C): a meta-analysis of the liraglutide development program. Endocr Pract. 2011 Nov-Dec;17(6):906-13. doi: 10.4158/ep.17.6.906. PMID 22193143
- [Result] Zinman B, Schmidt WE, Moses A, Lund N, Gough S. Achieving a clinically relevant composite outcome of an HbA1c of <7% without weight gain or hypoglycaemia in type 2 diabetes: a meta-analysis of the liraglutide clinical trial programme. Diabetes Obes Metab. 2012 Jan;14(1):77-82. doi: 10.1111/j.1463-1326.2011.01493.x. Epub 2011 Oct 30. PMID 21883806
- [Result] Davies MJ, Chubb BD, Smith IC, Valentine WJ. Cost-utility analysis of liraglutide compared with sulphonylurea or sitagliptin, all as add-on to metformin monotherapy in Type 2 diabetes mellitus. Diabet Med. 2012 Mar;29(3):313-20. doi: 10.1111/j.1464-5491.2011.03429.x. PMID 21883438
- [Result] Nauck M, Frid A, Hermansen K, Thomsen AB, During M, Shah N, Tankova T, Mitha I, Matthews DR. Long-term efficacy and safety comparison of liraglutide, glimepiride and placebo, all in combination with metformin in type 2 diabetes: 2-year results from the LEAD-2 study. Diabetes Obes Metab. 2013 Mar;15(3):204-12. doi: 10.1111/dom.12012. Epub 2012 Oct 11. PMID 22985213
- [Result] Niswender K, Pi-Sunyer X, Buse J, Jensen KH, Toft AD, Russell-Jones D, Zinman B. Weight change with liraglutide and comparator therapies: an analysis of seven phase 3 trials from the liraglutide diabetes development programme. Diabetes Obes Metab. 2013 Jan;15(1):42-54. doi: 10.1111/j.1463-1326.2012.01673.x. Epub 2012 Sep 9. PMID 22862847
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] King AB, Montanya E, Pratley RE, Blonde L, Svendsen CB, Donsmark M, Sesti G. Liraglutide achieves A1C targets more often than sitagliptin or exenatide when added to metformin in patients with type 2 diabetes and a baseline A1C <8.0%. Endocr Pract. 2013 Jan-Feb;19(1):64-72. doi: 10.4158/EP12232.OR. PMID 23186975
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Derived] Fonseca VA, Devries JH, Henry RR, Donsmark M, Thomsen HF, Plutzky J. Reductions in systolic blood pressure with liraglutide in patients with type 2 diabetes: insights from a patient-level pooled analysis of six randomized clinical trials. J Diabetes Complications. 2014 May-Jun;28(3):399-405. doi: 10.1016/j.jdiacomp.2014.01.009. Epub 2014 Jan 21. PMID 24561125
- [Derived] Hegedus L, Moses AC, Zdravkovic M, Le Thi T, Daniels GH. GLP-1 and calcitonin concentration in humans: lack of evidence of calcitonin release from sequential screening in over 5000 subjects with type 2 diabetes or nondiabetic obese subjects treated with the human GLP-1 analog, liraglutide. J Clin Endocrinol Metab. 2011 Mar;96(3):853-60. doi: 10.1210/jc.2010-2318. Epub 2011 Jan 5. PMID 21209033
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 170 centres in 21 countries: Argentina (4), Australia (19), Belgium (6), Bulgaria (1), Germany (33), Denmark (9), Spain (14), United Kingdom (11), Croatia (2), Hungary (5), Ireland (4), India (5), Italy (10), The Netherlands (5), New Zealand (3), Norway (8), Romania (3), Russia (6), Sweden (8), Slovakia (7) and South Africa (7)
Pre-assignment Details: Eligible subjects discontinued their oral anti-diabetic drug treatment and commenced a 3-week period of forced titration of metformin followed by a 3-week maintenance period. Subjects on current metformin therapy could go through a modified titration period or advance directly to the 3-week maintenance period at the discretion of the investigator.
Groups:
- Lira 0.6 + Met: Liraglutide 0.6 mg/day + glimepiride placebo + metformin 1.5-2.0 g/day, weeks 0-26 (double-blinded period) and open-label liraglutide 0.6 mg/day + metformin 1.5-2.0 g/day in the extension period (weeks 26-104)
- Lira 1.2 + Met: Liraglutide 1.2 mg/day + glimepiride placebo + metformin 1.5-2.0 g/day, weeks 0-26 (double-blinded period) and open-label liraglutide 1.2 mg/day + metformin 1.5-2.0 g/day in the extension period (weeks 26-104)
- Lira 1.8 + Met: Liraglutide 1.8 mg/day + glimepiride placebo + metformin 1.5-2.0 g/day, weeks 0-26 (double-blinded period) and open-label liraglutide 1.8 mg/day + metformin 1.5-2.0 g/day in the extension period (weeks 26-104)
- Met Mono: Metformin 1.5-2.0 g/day + liraglutide placebo + glimepiride placebo, weeks 0-26 (double-blinded period) and open-label metformin 1.5-2.0 g/day in the extension period (weeks 26-104)
- Met + Glim: Glimepiride 4 mg/day + metformin 1.5-2.0 g/day + liraglutide placebo, weeks 0-26 (double-blinded period) and open-label glimepiride 4 mg/day + metformin 1.5-2.0 g/day in the extension period (weeks 26-104)
Period: Double-Blind, 6 Months
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Started | 242 (Randomised) | 241 (Randomised) | 242 (Randomised) | 122 (Randomised) | 244 (Randomised)
Exposed to Study Drug | 242 | 240 (Subject withdrew before exposure to drug, and thus not included in the safety and ITT analysis sets) | 242 | 121 (Subject withdrew before exposure to drug, and thus not included in the safety and ITT analysis sets) | 242 (Subjects withdrew before exposure to drug, and thus not included in the safety and ITT analysis sets)
Completed | 208 | 197 | 191 | 74 | 210
Not Completed | 34 | 44 | 51 | 48 | 34
Not completed — Adverse Event | 11 | 23 | 29 | 2 | 8
Not completed — Lack of Efficacy | 19 | 8 | 13 | 29 | 9
Not completed — Protocol Violation | 2 | 4 | 4 | 4 | 5
Not completed — Lost to follow up | 0 | 1 | 0 | 0 | 0
Not completed — Poor compliance/Non-compliance | 0 | 1 | 0 | 0 | 0
Not completed — Consent withdrawn | 0 | 3 | 4 | 10 | 4
Not completed — Subject decision/No wish to continue | 0 | 2 | 1 | 0 | 2
Not completed — Move | 0 | 1 | 0 | 0 | 0
Not completed — Tendency to low blood glucose levels | 0 | 0 | 0 | 0 | 1
Not completed — FPG exceeds limits/too high | 1 | 0 | 0 | 2 | 0
Not completed — Work commitment | 0 | 0 | 0 | 0 | 1
Not completed — Investigator decision | 0 | 0 | 0 | 0 | 1
Not completed — Lack of time | 1 | 0 | 0 | 0 | 0
Not completed — Hypoglycaemia/Hypoglycemia | 0 | 0 | 0 | 0 | 2
Not completed — Hyperglicaemia | 0 | 0 | 0 | 1 | 0
Not completed — metformin titrated <1500 mg or >2000 mg | 0 | 0 | 0 | 0 | 1
Not completed — Fear of experiencing AE again | 0 | 1 | 0 | 0 | 0
Period: Open-Label Extension, 18 Months
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Started | 208 | 197 | 191 | 74 | 210
Completed | 130 | 137 | 118 | 31 | 113
Not Completed | 78 | 60 | 73 | 43 | 97
Not completed — Withdrawals between 6 and 24 months | 19 | 14 | 27 | 11 | 22
Not completed — Adverse Event | 11 | 8 | 6 | 1 | 6
Not completed — Lack of Efficacy | 41 | 33 | 37 | 27 | 63
Not completed — Protocol Violation | 7 | 5 | 3 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim | Total
Number analyzed (Participants) | 242 | 240 | 242 | 121 | 242 | 1087
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (10.5) | 57.2 (9.2) | 56.8 (9.4) | 56.0 (9.4) | 57.3 (8.8) | 56.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 111 | 100 | 49 | 103 | 454
  Male | 151 | 129 | 142 | 72 | 139 | 633
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 31 | 19 | 18 | 9 | 21 | 98
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 9 | 5 | 3 | 5 | 26
  White | 202 | 210 | 214 | 106 | 214 | 946
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 5 | 3 | 2 | 17
Previous anti-diabetic treatment [Number; unit: participants]
  Mono-therapy | 81 | 90 | 82 | 41 | 90 | 384
  Combination therapy | 161 | 150 | 160 | 80 | 152 | 703
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 30.5 (4.8) | 31.1 (4.8) | 30.9 (4.6) | 31.6 (4.4) | 31.2 (4.6) | 31.0 (4.7)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis of diabetes
  years | 7.0 (4.8) | 6.8 (4.9) | 7.8 (5.2) | 7.9 (6.0) | 7.7 (5.3) | 7.4 (5.2)
HbA1c [Mean (Standard Deviation); unit: percentage of total haemoglobin] — Glycosylated Haemoglobin at screening
  percentage of total haemoglobin | 8.4 (0.9) | 8.3 (0.9) | 8.3 (0.9) | 8.4 (1.0) | 8.4 (0.9) | 8.4 (0.9)
Height [Mean (Standard Deviation); unit: m] | 1.69 (0.10) | 1.68 (0.11) | 1.69 (0.10) | 1.69 (0.10) | 1.69 (0.11) | 1.69 (0.10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated A1c (HbA1c) at Week 26
Description: Percentage point change in Glycosylated A1c (HbA1c) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: Intention to treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects who had been exposed to at least one dose of the study products.
Measure: Least Squares Mean (Standard Error); unit: Percentage point of total HbA1c
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 239 | 232 | 236 | 120 | 234
Percentage point of total HbA1c | -0.69 (0.07) | -0.97 (0.07) | -1.00 (0.07) | 0.09 (0.09) | -0.98 (0.07)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in HbA1c from baseline to end of treatment at 26 weeks was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline glycosylated A1c (HbA1c) as covariate; Test type: Non-Inferiority or Equivalence — Hypothesis testing was done in a hierarchical manner. First, it was tested whether liraglutide 1.8 mg+metformin was superior to placebo + metformin. Superiority was always concluded if the upper limit of the 2-sided 95% CI for the treatment difference was below 0%; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.09, 95% CI [-1.30 to -0.88]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Hypothesis testing was done in a hierarchical manner. As superiority of liraglutide 1.8 mg + metformin to metformin monotherapy was established, it was investigated whether liraglutide 1.8 mg + metformin was non-inferior to glimepiride + metformin. Non-inferiority was concluded if the upper limit of the 2-sided 95% CI for the treatment difference was below 0.4%; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -0.02, 95% CI [-0.19 to 0.15]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Hypothesis testing was done in a hierarchical manner. First, it was tested whether liraglutide 1.2 mg+metformin was superior to placebo + metformin. Superiority was always concluded if the upper limit of the 2-sided 95% CI for the treatment difference was below 0%; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.06, 95% CI [-1.27 to -0.85]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Hypothesis testing was done in a hierarchical manner. As superiority of liraglutide 1.2 mg + metformin to metformin monotherapy was established, it was investigated whether liraglutide 1.2 mg + metformin was non-inferior to glimepiride + metformin. Non-inferiority was concluded if the upper limit of the 2-sided 95% CI for the treatment difference was below 0.4%; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = 0.01, 95% CI [-0.16 to 0.18]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Hypothesis testing was done in a hierarchical manner. First, it was tested whether liraglutide 0.6 mg+metformin was superior to placebo + metformin. Superiority was always concluded if the upper limit of the 2-sided 95% CI for the treatment difference was below 0%; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -0.78, 95% CI [-0.99 to -0.57]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Hypothesis testing was done in a hierarchical manner. As superiority of liraglutide 0.6 mg + metformin to metformin monotherapy was established, it was investigated whether liraglutide 0.6 mg + metformin was non-inferior to glimepiride + metformin. Non-inferiority was concluded if the upper limit of the 2-sided 95% CI for the treatment difference was below 0.4%; p = 0.1026, ANCOVA; Estimated treatment difference, LS Mean = 0.29, 95% CI [0.12 to 0.46]
Statistical Analysis 7: Comparison: Met Mono vs Met + Glim; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — A test for superiority of glimepiride+metformin to metformin was performed to verify assay sensitivity. Superiority was always concluded if the upper limit of the 2-sided 95% CI for the treatment difference was below 0%; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.07, 95% CI [-1.28 to -0.86]

2. Secondary Outcome: Change in Body Weight at Week 26
Description: Change in body weight from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 242 | 236 | 241 | 121 | 237
kg | -1.78 (0.23) | -2.58 (0.24) | -2.79 (0.23) | -1.51 (0.31) | 0.95 (0.23)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in body weight from baseline to end of treatment at 26 weeks was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline body weight as covariate; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.8 mg + metformin and placebo + metfomine was calculated. If the upper limit of the 95% CI was below 0%, it was concluded that the given dose of liraglutide in combination with metformin was better than the comparator therapy; p = 0.0016, ANCOVA; Estimated treatment difference, LS Mean = -1.29, 95% CI [-2.16 to -0.41]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.8 mg + metformin and glimepiride + metfomine was calculated. If the upper limit of the 95% CI was below 0%, it was concluded that the given dose of liraglutide in combination with metformin was better than the comparator therapy; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -3.75, 95% CI [-4.48 to -3.01]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.2 mg + metformin and placebo + metfomine was calculated. If the upper limit of the 95% CI was below 0%, it was concluded that the given dose of liraglutide in combination with metformin was better than the comparator therapy; p = 0.0117, ANCOVA; Estimated treatment difference, LS Mean = -1.07, 95% CI [-1.94 to -0.19]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.2 mg + metformin and glimepirde + metfomine was calculated. If the upper limit of the 95% CI was below 0%, it was concluded that the given dose of liraglutide in combination with metformin was better than the comparator therapy; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -3.53, 95% CI [-4.27 to -2.79]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 0.6 mg + metformin and placebo + metfomine was calculated. If the upper limit of the 95% CI was below 0%, it was concluded that the given dose of liraglutide in combination with metformin was better than the comparator therapy; p = 0.8198, ANCOVA; Estimated treatment difference, LS Mean = -0.28, 95% CI [-1.15 to 0.60]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 0.6 mg + metformin and glimepirde + metfomine was calculated. If the upper limit of the 95% CI was below 0%, it was concluded that the given dose of liraglutide in combination with metformin was better than the comparator therapy; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -2.73, 95% CI [-3.47 to -2.00]

3. Secondary Outcome: Change in Body Weight at Week 104
Description: Change in body weight from baseline (week 0) to 104 weeks (end of treatment)
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 242 | 236 | 241 | 121 | 237
kg | -2.07 (0.28) | -3.03 (0.29) | -2.91 (0.28) | -1.80 (0.38) | 0.70 (0.29)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in body weight from baseline to end of treatment at 104 weeks was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline body weight as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0378, ANCOVA; Estimated treatment difference, LS Mean = -1.11, 95% CI [-2.18 to -0.05]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -3.61, 95% CI [-4.51 to -2.72]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p = 0.0185, ANCOVA; Estimated treatment difference, LS Mean = -1.23, 95% CI [-2.30 to -0.16]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -3.73, 95% CI [-4.64 to -2.83]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p = 0.9069, ANCOVA; Estimated treatment difference, LS Mean = -0.27, 95% CI [-1.33 to 0.80]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -2.77, 95% CI [-3.67 to -1.87]

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) at Week 26
Description: Change in fasting plasma glucose (FPG) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 238 | 234 | 235 | 116 | 234
mmol/L | -1.13 (0.15) | -1.63 (0.16) | -1.68 (0.15) | 0.40 (0.21) | -1.31 (0.16)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in fasting plasma glucose from baseline to end of treatment at 26 weeks was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline fasting plasma glucose as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -2.09, 95% CI [-2.68 to -1.50]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.1845, ANCOVA; Estimated treatment difference, LS Mean = -0.38, 95% CI [-0.87 to 0.11]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -2.04, 95% CI [-2.63 to -1.44]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; Change in fasting plasma glucose from baseline to end of treatment at 26 weeks was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline fasting plasma glucose t as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p = 0.3047, ANCOVA; Estimated treatment difference, LS Mean = -0.33, 95% CI [-0.82 to 0.17]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.53, 95% CI [-2.12 to -0.94]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p = 0.8079, ANCOVA; Estimated treatment difference, LS Mean = 0.18, 95% CI [-0.32 to 0.67]

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) at Week 104
Description: Change in Fasting plasma glucose (FPG) from baseline (week 0) to 104 weeks (end of treatment)
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 238 | 233 | 234 | 116 | 234
mmol/L | -0.80 (0.17) | -1.20 (0.18) | -1.18 (0.17) | 0.75 (0.23) | -0.64 (0.17)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in fasting plasma glucose from baseline to end of treatment at 104 weeks was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline fasting plasma glucose as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.93, 95% CI [-2.58 to -1.28]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.0542, ANCOVA; Estimated treatment difference, LS Mean = -0.53, 95% CI [-1.08 to 0.01]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.95, 95% CI [-2.60 to -1.30]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; Change in fasting plasma glucose from baseline to end of treatment at 104 weeks was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline fasting plasma glucose t as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p = 0.0451, ANCOVA; Estimated treatment difference, LS Mean = -0.55, 95% CI [-1.10 to -0.01]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.55, 95% CI [-2.20 to -0.90]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p = 0.9006, ANCOVA; Estimated treatment difference, LS Mean = -0.15, 95% CI [-0.70 to 0.39]

6. Secondary Outcome: Change in Mean Prandial Increments of Plasma Glucose Based on Self-measured 7-point Plasma Glucose Profiles at Week 26
Description: Change in mean prandial increments of plasma glucose based on self-measured 7-point plasma glucose profiles from baseline (week 0) to 26 weeks (end of randomisation). The 7 time points for self-measurements were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner) and at bedtime.
  Mean prandial increments of plasma glucose were calculated as the sum of the plasma glucose differences between values measured before and after a meal (breakfast, lunch and dinner) divided by three.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/l
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 214 | 207 | 205 | 90 | 213
mmol/l | -0.23 (0.12) | -0.40 (0.13) | -0.56 (0.12) | -0.44 (0.18) | -0.44 (0.12)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in prandial increments of plasma glucose from baseline to 26 weeks of treatment was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.8871, ANCOVA; Estimated treatment difference, LS Mean = -0.13, 95% CI [-0.62 to 0.36]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.8695, ANCOVA; Estimated treatment difference, LS Mean = -0.12, 95% CI [-0.51 to 0.27]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p = 0.9994, ANCOVA; Estimated treatment difference, LS Mean = 0.03, 95% CI [-0.46 to 0.52]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p = 0.9984, ANCOVA; Estimated treatment difference, LS Mean = 0.04, 95% CI [-0.35 to 0.43]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; Change in mean prandial increments of plasma glucose from baseline to 26 weeks of treatment was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p = 0.6201, ANCOVA; Estimated treatment difference, LS Mean = 0.21, 95% CI [-0.28 to 0.70]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 6, analysis 5]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p = 0.4831, ANCOVA; Estimated treatment difference, LS Mean = 0.21, 95% CI [-0.18 to 0.60]

7. Primary Outcome: Change in Glycosylated A1c (HbA1c) at Week 104
Description: Change in glycosylated A1c (HbA1c) baseline (week 0) to 104 weeks (end of randomisation)
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total haemoglobin
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 239 | 231 | 235 | 120 | 234
percentage of total haemoglobin | -0.36 (0.08) | -0.56 (0.08) | -0.58 (0.08) | 0.25 (0.10) | -0.50 (0.08)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in HbA1c from baseline to end of treatment at 104 weeks was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline glycosylated A1c (HbA1c) as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -0.83, 95% CI [-1.07 to -0.59]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -0.08, 95% CI [-0.28 to 0.12]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; Change in HbA1c from baseline to end of treatment was at 104 weeks analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline glycosylated A1c (HbA1c) as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -0.81, 95% CI [-1.05 to -0.57]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 4]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -0.07, 95% CI [-0.27 to 0.13]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 5]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -0.61, 95% CI [-0.85 to -0.37]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 6]; p = 0.0052, ANCOVA; Estimated treatment difference, LS Mean = 0.14, 95% CI [-0.06 to 0.34]
Statistical Analysis 7: Comparison: Met Mono vs Met + Glim; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — A test for superiority of glimepiride+metformin to placebo metformin was performed to verify assay sensitivity. Superiority was always concluded if the upper limit of the 2-sided 95% CI for the treatment difference was below 0%; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -0.75, 95% CI [-0.99 to -0.51]

8. Secondary Outcome: Change in Mean Prandial Increments of Plasma Glucose Based on Self-measured 7-point Plasma Glucose Profiles at Week 104
Description: Change in mean prandial increments of plasma glucose based on self-measured 7-point plasma glucose profiles from baseline (week 0) to 104 weeks (end of treatment). The 7 time points for self-measurements were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner) and at bedtime.
  Mean prandial increments of plasma glucose were calculated as the sum of the plasma glucose differences between values measured before and after a meal (breakfast, lunch and dinner) divided by three.
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 218 | 208 | 206 | 90 | 215
mmol/L | -0.27 (0.12) | -0.56 (0.13) | -0.44 (0.13) | -0.20 (0.18) | -0.29 (0.13)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in prandial increments of plasma glucose from baseline to 104 weeks of treatment was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.5282, ANCOVA; Estimated treatment difference, LS Mean = -0.24, 95% CI [-0.74 to 0.26]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.7644, ANCOVA; Estimated treatment difference, LS Mean = -0.15, 95% CI [-0.55 to 0.25]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p = 0.2063, ANCOVA; Estimated treatment difference, LS Mean = -0.36, 95% CI [-0.86 to 0.14]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p = 0.2678, ANCOVA; Estimated treatment difference, LS Mean = -0.28, 95% CI [-0.68 to 0.12]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p = 0.9887, ANCOVA; Estimated treatment difference, LS Mean = -0.07, 95% CI [-0.57 to 0.43]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p = 0.9998, ANCOVA; Estimated treatment difference, LS Mean = 0.02, 95% CI [-0.38 to 0.42]

9. Secondary Outcome: Change in Mean Post Prandial Plasma Glucose Based on Self-measured 7-point Plasma Glucose Profiles at Week 26
Description: Change in mean post prandial plasma glucose from baseline (Week 0) to 26 weeks (end of randomisation). The 7 time points for self-measurements were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner) and at bedtime. Mean post prandial plasma glucose were calculated as the sum of the post pradial plasma glucose values divided by three.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 214 | 207 | 205 | 90 | 214
mmol/L | -1.68 (0.16) | -2.33 (0.17) | -2.57 (0.16) | -0.62 (0.24) | -2.46 (0.16)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in post prandial increments of plasma glucose from baseline to 26 weeks of treatment was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.95, 95% CI [-2.60 to -1.30]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.9670, ANCOVA; Estimated treatment difference, LS Mean = -0.11, 95% CI [-0.62 to 0.41]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.72, 95% CI [-2.36 to -1.07]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p = 0.9368, ANCOVA; Estimated treatment difference, LS Mean = 0.13, 95% CI [-0.39 to 0.64]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p = 0.0003, ANCOVA; Estimated treatment difference, LS Mean = -1.06, 95% CI [-1.71 to -0.42]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p = 0.0008, ANCOVA; Estimated treatment difference, LS Mean = 0.78, 95% CI [0.27 to 1.29]

10. Secondary Outcome: Change in Mean Post Prandial Plasma Glucose Based on Self-measured 7-point Plasma Glucose Profiles at Week 104
Description: Change in mean post prandial plasma glucose from baseline (Week 0) to 104 weeks (end of treatment) The 7 time points for self-measurements were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner) and at bedtime. Mean post prandial plasma glucose were calculated as the sum of the post pradial plasma glucose values divided by three.
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 218 | 208 | 206 | 90 | 216
mmol/L | -1.59 (0.18) | -2.22 (0.18) | -2.10 (0.18) | -0.43 (0.26) | -1.80 (0.18)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in post prandial increments of plasma glucose from baseline to 104 weeks of treatment was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.66, 95% CI [-2.37 to -0.96]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 10, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.5048, ANCOVA; Estimated treatment difference, LS Mean = -0.30, 95% CI [-0.86 to 0.26]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 10, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.0001, ANCOVA; Estimated treatment difference, LS Mean = -1.79, 95% CI [-2.49 to -1.08]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 10, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p = 0.2005, ANCOVA; Estimated treatment difference, LS Mean = -0.42, 95% CI [-0.98 to 0.14]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 10, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p = 0.0003, ANCOVA; Estimated treatment difference, LS Mean = -1.16, 95% CI [-1.86 to -0.46]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 10, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p = 0.7871, ANCOVA; Estimated treatment difference, LS Mean = 0.21, 95% CI [-0.35 to 0.76]

11. Secondary Outcome: Change in Beta-cell Function at Week 26
Description: Change in beta cell function from baseline (week 0) to 16 weeks (end of treatment). Beta-cell function was derived from fasting plasma glucose (FPG) and fasting insulin concentrations using the homeostasic model assessment (HOMA) method which uses the assumption that normal-weight normal subjects aged under 35 years have a 100% beta-cell function (HOMA-B).
  Beta-cell function: HOMA-B (%) = 20∙fasting insulin[uU/mL] divided by (FPG mmol/L]-3.5).
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point (%point)
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 229 | 224 | 224 | 109 | 226
percentage point (%point) | 20.45 (5.19) | 20.33 (5.34) | 26.12 (5.20) | -1.63 (7.19) | 24.68 (5.25)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in HOMA-B from baseline to 26 weeks of treatment was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0031, ANCOVA; Estimated treatment difference, LS Mean = 27.75, 95% CI [7.83 to 47.67]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 11, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.9987, ANCOVA; Estimated treatment difference, LS Mean = 1.44, 95% CI [-15.03 to 17.90]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 11, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p = 0.0263, ANCOVA; Estimated treatment difference, LS Mean = 21.96, 95% CI [2.04 to 41.87]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 11, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p = 0.9227, ANCOVA; Estimated treatment difference, LS Mean = -4.36, 95% CI [-20.94 to 12.22]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 11, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p = 0.0253, ANCOVA; Estimated treatment difference, LS Mean = 22.08, 95% CI [2.15 to 42.01]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 11, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p = 0.9293, ANCOVA; Estimated treatment difference, LS Mean = -4.23, 95% CI [-20.78 to 12.31]

12. Secondary Outcome: Change in Beta-cell Function at Week 104
Description: as for outcome 11
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point (%point)
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 230 | 224 | 224 | 110 | 226
percentage point (%point) | 64.48 (24.93) | 27.30 (25.70) | 17.81 (25.03) | -7.89 (34.47) | 11.25 (25.27)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Met Mono; Change in HOMA-B from baseline to 104 weeks of treatment was analyzed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.8821, ANCOVA; Estimated treatment difference, LS Mean = 25.71, 95% CI [-69.84 to 121.26]
Statistical Analysis 2: Comparison: Lira 1.8 + Met vs Met + Glim; [analysis description as in outcome 12, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.9989, ANCOVA; Estimated treatment difference, LS Mean = 6.56, 95% CI [-72.66 to 85.79]
Statistical Analysis 3: Comparison: Lira 1.2 + Met vs Met Mono; [analysis description as in outcome 12, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p = 0.7292, ANCOVA; Estimated treatment difference, LS Mean = 35.20, 95% CI [-60.33 to 130.72]
Statistical Analysis 4: Comparison: Lira 1.2 + Met vs Met + Glim; [analysis description as in outcome 12, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 4]; p = 0.9689, ANCOVA; Estimated treatment difference, LS Mean = 16.05, 95% CI [-63.69 to 95.79]
Statistical Analysis 5: Comparison: Lira 0.6 + Met vs Met Mono; [analysis description as in outcome 12, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 5]; p = 0.1818, ANCOVA; Estimated treatment difference, LS Mean = 72.38, 95% CI [-23.15 to 167.90]
Statistical Analysis 6: Comparison: Lira 0.6 + Met vs Met + Glim; [analysis description as in outcome 12, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 6]; p = 0.2978, ANCOVA; Estimated treatment difference, LS Mean = 53.23, 95% CI [-26.30 to 132.76]

13. Secondary Outcome: Hypoglycaemic Episodes at Week 26
Description: Total number of hypoglycaemic episodes occuring after baseline (week 0) until week 26 (end of randomisation). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: weeks 0-26
Population: Safety analysis set is all randomised subjects who were exposed to at least one dose of study product.
Measure: Number; unit: episodes
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 242 | 240 | 242 | 121 | 242
episodes
  Major | 0 | 0 | 0 | 0 | 0
  Minor | 15 | 3 | 9 | 6 | 136
  Symptoms only | 17 | 7 | 22 | 10 | 175

14. Secondary Outcome: Hypoglycaemic Episodes at Week 104
Description: Total number of hypoglycaemic episodes occuring after baseline (week 0) until 104 weeks (end of treatment). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: weeks 0-104
Population: Safety analysis set is all randomised subjects who were exposed to at least one dose of study product.
Measure: Number; unit: episodes
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Number analyzed (Participants) | 242 | 240 | 242 | 121 | 242
episodes
  All | 52 | 51 | 49 | 18 | 524
  Major | 0 | 1 | 0 | 0 | 0
  Minor | 23 | 26 | 22 | 6 | 284
  Symptoms only | 29 | 24 | 27 | 12 | 240

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 24 months of treatment
Description: The safety analysis set is all randomised subjects who were exposed to at least one dose of study product.
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Met Mono | Met + Glim
Serious Adverse Events (participants affected / at risk) | 36/242 | 25/240 | 16/242 | 9/121 | 24/242
Other Adverse Events (participants affected / at risk) | 132/242 | 144/240 | 158/242 | 44/121 | 128/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 0.6 + Met (N=242) | Lira 1.2 + Met (N=240) | Lira 1.8 + Met (N=242) | Met Mono (N=121) | Met + Glim (N=242)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sympathetic nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess sweat gland (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant lymphoma unclassifiable high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral hypoperfusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcitonin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial stenosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 0.6 + Met (N=242) | Lira 1.2 + Met (N=240) | Lira 1.8 + Met (N=242) | Met Mono (N=121) | Met + Glim (N=242)
Nasopharyngitis (Infections and infestations) | 43 (69) | 36 (70) | 36 (43) | 12 (21) | 49 (80)
Influenza (Infections and infestations) | 14 (17) | 15 (18) | 17 (27) | 5 (6) | 18 (27)
Upper respiratory tract infection (Infections and infestations) | 11 (16) | 14 (19) | 15 (19) | 4 (6) | 12 (19)
Bronchitis (Infections and infestations) | 10 (10) | 13 (16) | 12 (13) | 3 (3) | 15 (20)
Nausea (Gastrointestinal disorders) | 30 (33) | 42 (50) | 52 (70) | 5 (6) | 10 (14)
Diarrhoea (Gastrointestinal disorders) | 31 (40) | 27 (43) | 40 (50) | 5 (5) | 14 (20)
Vomiting (Gastrointestinal disorders) | 19 (21) | 18 (22) | 24 (26) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 12 (13) | 6 (6) | 22 (27) | 1 (4) | 7 (11)
Gastritis (Gastrointestinal disorders) | 10 (11) | 8 (11) | 13 (13) | 1 (1) | 4 (6)
Toothache (Gastrointestinal disorders) | 6 (6) | 13 (14) | 7 (8) | 6 (8) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (21) | 15 (17) | 17 (20) | 5 (6) | 21 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 5 (5) | 9 (12) | 5 (7) | 19 (22)
Headache (Nervous system disorders) | 26 (41) | 34 (40) | 35 (51) | 8 (8) | 32 (55)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 10 (10) | 15 (17) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 14 (15) | 10 (10) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 11 (11) | 13 (15) | 11 (11) | 2 (2) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (6) | 2 (3) | 2 (2) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.